CLINICAL TRIAL: NCT02585206
Title: Optimizing Text Messaging to Improve Adherence to Web-Based Cessation Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Truth Initiative (Other)
Responsible Party: Principal Investigator, Amanda L. Graham, PhD, Director, Research Development, Truth Initiative
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01DA038139 (NIH)
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Smoking Cessation
Keywords: Mobile Phone; Text Messaging; Internet; Tobacco Use
MeSH Terms: conditions — Smoking Cessation; Tobacco Use

STUDY DESIGN:
Intervention Model Description: Phase I: full factorial design of four factors each with 2 levels (16 arms); Phase II: 2-arm randomized trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- Arm 1 (No Intervention): All 4 factors off - standard text message program
  Personalization OFF Integration OFF Dynamic Tailoring OFF Message Intensity OFF
- Arm 2 (Active Comparator): Personalization OFF Integration OFF Dynamic Tailoring OFF Message Intensity ON
  Interventions: Behavioral: Message Intensity
- Arm 3 (Active Comparator): Personalization OFF Integration OFF Dynamic Tailoring ON Message Intensity OFF
  Interventions: Behavioral: Dynamic Tailoring
- Arm 4 (Active Comparator): Personalization OFF Integration OFF Dynamic Tailoring ON Message Intensity ON
  Interventions: Behavioral: Dynamic Tailoring; Behavioral: Message Intensity
- Arm 5 (Active Comparator): Personalization OFF Integration ON Dynamic Tailoring OFF Message Intensity OFF
  Interventions: Behavioral: Integration
- Arm 6 (Active Comparator): Personalization OFF Integration ON Dynamic Tailoring OFF Message Intensity ON
  Interventions: Behavioral: Integration; Behavioral: Message Intensity
- Arm 7 (Active Comparator): Personalization OFF Integration ON Dynamic Tailoring ON Message Intensity OFF
  Interventions: Behavioral: Integration; Behavioral: Dynamic Tailoring
- Arm 8 (Active Comparator): Personalization OFF Integration ON Dynamic Tailoring ON Message Intensity ON
  Interventions: Behavioral: Integration; Behavioral: Dynamic Tailoring; Behavioral: Message Intensity
- Arm 9 (Active Comparator): Personalization ON Integration OFF Dynamic Tailoring OFF Message Intensity OFF
  Interventions: Behavioral: Personalization
- Arm 10 (Active Comparator): Personalization ON Integration OFF Dynamic Tailoring OFF Message Intensity ON
  Interventions: Behavioral: Personalization; Behavioral: Message Intensity
- Arm 11 (Active Comparator): Personalization ON Integration OFF Dynamic Tailoring ON Message Intensity OFF
  Interventions: Behavioral: Personalization; Behavioral: Dynamic Tailoring
- Arm 12 (Active Comparator): Personalization ON Integration OFF Dynamic Tailoring ON Message Intensity ON
  Interventions: Behavioral: Personalization; Behavioral: Dynamic Tailoring; Behavioral: Message Intensity
- Arm 13 (Active Comparator): Personalization ON Integration ON Dynamic Tailoring OFF Message Intensity OFF
  Interventions: Behavioral: Personalization; Behavioral: Integration
- Arm 14 (Active Comparator): Personalization ON Integration ON Dynamic Tailoring OFF Message Intensity ON
  Interventions: Behavioral: Personalization; Behavioral: Integration; Behavioral: Message Intensity
- Arm 15 (Active Comparator): Personalization ON Integration ON Dynamic Tailoring ON Message Intensity OFF
  Interventions: Behavioral: Personalization; Behavioral: Integration; Behavioral: Dynamic Tailoring
- Arm 16 (Active Comparator): Personalization ON Integration ON Dynamic Tailoring ON Message Intensity ON
  Interventions: Behavioral: Personalization; Behavioral: Integration; Behavioral: Dynamic Tailoring; Behavioral: Message Intensity
- WEB (No Intervention): Phase II arm.
  Full access to standard BecomeAnEX.org web-based smoking cessation program.
- WEB+OA_TXT (Active Comparator): Phase II arm.
  Full access to standard BecomeAnEX.org web-based smoking cessation program PLUS optimal-adherence text message program from Phase I.
  Interventions: Behavioral: Optimal-Adherence Text

INTERVENTIONS:
Behavioral: Personalization — Phase I Factor
  Personalized text messages using the participant's username and gender ("Check out the EX Community for tips/support from other men who have quit. They've been there and can help you do this, QuitForever!"). Both data points will be pulled from BecomeAnEX registration data.
  Arms: Arm 10; Arm 11; Arm 12; Arm 13; Arm 14; Arm 15; Arm 16; Arm 9
Behavioral: Integration — Phase I Factor
  Interactive messages to facilitate engagement via text with the 6 interactive intervention components of the BecomeAnEX web intervention:
  Set your quit date Cigarette tracker Beat your smoking triggers Build your support system Choose a quit smoking aid Community
  Integration will allow interaction with the web-based program via text message; for example, when a user sets a quit date via the website, it will trigger text messages tailored to the quit date; likewise, if a user sets a quit date via the text system, it will be populated in the website and drive the user experience online.
  Arms: Arm 13; Arm 14; Arm 15; Arm 16; Arm 5; Arm 6; Arm 7; Arm 8
Behavioral: Dynamic Tailoring — Individually tailored message to remind/reinforce users about BecomeAnEX information/tools they have already used, or to prompt users to take actions they have not yet taken.
  Arms: Arm 11; Arm 12; Arm 15; Arm 16; Arm 3; Arm 4; Arm 7; Arm 8
Behavioral: Message Intensity — Phase I Factor
  Varying levels of text message intensity over a 12-week period.
  Arms: Arm 10; Arm 12; Arm 14; Arm 16; Arm 2; Arm 4; Arm 6; Arm 8
Behavioral: Optimal-Adherence Text — Optimal-adherence text message intervention developed in Phase I
  Other Names: OA_TXT
  Arms: WEB+OA_TXT

SUMMARY:
This study is comprised of 2 phases to study the impact of a text message system on overall adherence to a web-based smoking cessation program. Phase I uses a full factorial design to identify the most optimal text message intervention to maximize adherence to the BecomeAnEX.org smoking cessation program. Phase II is a randomized controlled trial that compares regular BecomeAnEX users to those who will receive the optimized text message intervention (from Phase I) in conjunction with BecomeAnEX for impact on long-term abstinence.

DETAILED DESCRIPTION:
This study is comprised of 2 active phases, all conducted with registered users on BecomeAnEX.org, a well-established smoking cessation website.

Phase I involves the initial development and optimization of the text message intervention. The investigators will examine the impact of 4 experimental text message intervention features on smokers' adherence to a web-based cessation intervention during the first 3 months of program enrollment. The investigators will utilize a full factorial design where participants will be randomized to 1 of 2 levels of each of the following features: 1) personalization (yes/no), 2) integration (yes/no), 3) dynamic tailoring (yes/no), and 4) message intensity (standard vs. decreasing). The primary outcome in Phase I will be a composite metric of utilization.

Phase II involves a 2-arm randomized trial that compares WEB alone to WEB plus the text message intervention from Phase I that yields optimal adherence (WEB+OA_TXT). The randomized trial will use a repeated measures design, with assessments at baseline, 3, 9, and 15 months. Follow-ups at 3, 9, and 15 months correspond to 0, 6, and 12 months post-treatment. The primary outcome is 30-day point prevalence abstinence (ppa) at 9-months. The investigators will assess and validate smoking status at all follow-ups. Other outcomes include motivation to quit, quit attempts, and continuous abstinence.

ELIGIBILITY:
Inclusion Criteria:

* US residency
* Current smoker
* Access to and willingness to receive text messages on a mobile phone
* Access to Internet
* Access to and willingness to receive email communication from study personnel

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1485 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Phase I - Composite adherence metric | 3 months
  The investigators will create a composite metric of adherence for each Phase I participant using a weighted sum of their total number of number of visits, as well as of their page views, time on site, and use of the 6 interactive components of the site per visit during 3 months post-enrollment.
Phase II - 30-day point prevalence abstinence | 9 months post randomization
  Self-reported 30-day point prevalence abstinence at 9 months post randomization

SECONDARY OUTCOMES:
Phase II - 30day point prevalence abstinence | 3 months post randomization
  Self-reported 30-day point prevalence abstinence at 3 months post randomization
Phase II - 30day point prevalence abstinence | 15 months post randomization
  Self-reported 30-day point prevalence abstinence at 15 months post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Amanda L Graham, PhD, Principal Investigator — Truth Initiative
Locations (1):
- Truth Initiative, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Graham AL, Jacobs MA, Cohn AM, Cha S, Abroms LC, Papandonatos GD, Whittaker R. Optimising text messaging to improve adherence to web-based smoking cessation treatment: a randomised control trial protocol. BMJ Open. 2016 Mar 30;6(3):e010687. doi: 10.1136/bmjopen-2015-010687. PMID 27029775
- [Derived] Graham AL, Papandonatos GD, Cha S, Amato MS, Jacobs MA, Cohn AM, Abroms LC, Whittaker R. Effectiveness of an optimized text message and Internet intervention for smoking cessation: A randomized controlled trial. Addiction. 2022 Apr;117(4):1035-1046. doi: 10.1111/add.15677. Epub 2021 Sep 28. PMID 34472676
- [Derived] Graham AL, Papandonatos GD, Jacobs MA, Amato MS, Cha S, Cohn AM, Abroms LC, Whittaker R. Optimizing Text Messages to Promote Engagement With Internet Smoking Cessation Treatment: Results From a Factorial Screening Experiment. J Med Internet Res. 2020 Apr 2;22(4):e17734. doi: 10.2196/17734. PMID 32238338